CLINICAL TRIAL: NCT03551990
Title: Influence of Motor Proteins on Muscle Atrophy in Cancer Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EMS Tumor Motor Proteins
Record Dates: First submitted 2017-05-10; First posted 2018-06-11 (Actual); Last update posted 2018-06-11 (Actual); Status verified 2018-05

CONDITIONS: Cancer; Muscle Atrophy
Keywords: Whole-body electromyostimulation; WB-EMS; Cancer; Muscle atrophy; Muscle protein; Exercise; Muscle fiber
MeSH Terms: conditions — Neoplasms; Muscular Atrophy; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group; patients without a tumor disease, surgery (No Intervention): Control group with patients without a tumor disease but with indication for surgery in close proximity to the M. rectus abdominis
- Control group; tumor patients, surgery (No Intervention): Control group with patients with solid tumors; patients with pancreatic, colorectal, esophageal, gastric and liver solid tumors with indication for surgery in close proximity to the M. rectus abdominis
- Intervention group; tumor patients, WB-EMS, surgery (Experimental): Intervention group with patients with solid tumors who do perform an 8-week physical training in form of whole-body electromyostimulation (WB-EMS); patients with pancreatic, colorectal, esophageal, gastric and liver solid tumors with indication for surgery in close proximity to the M. rectus abdominis
  Interventions: Procedure: whole-body electromyostimulation WB-EMS

INTERVENTIONS:
Procedure: whole-body electromyostimulation WB-EMS — Patients of the WB-EMS group will perform whole-body electromyostimulation (WB-EMS) training sessions twice a week over a period of 8 weeks. To allow muscle recovery a break of at least 2 days between the sessions will be scheduled. To adapt the patients to the WB-EMS intervention, the training duration will be gradually increased (week 1, 12 min; increase of 2 min/week; week 5-8, 20 min). WB-EMS training sessions will include light physical exercises according to a video tutorial and individually supervised by certified physio therapists.
  Arms: Intervention group; tumor patients, WB-EMS, surgery

SUMMARY:
The aim of the study is to investigate the effect of exercise in form of whole-body electromyostimulation (WB-EMS) on early tumor-induced muscular dysfunction. It is anticipated to gain detailed knowledge about composition and metabolism of skeletal muscle cells, and single muscle fiber functionality. To determine key factors leading to impaired force generation and thus decreased muscle strength in cancer patients who are suspected to develop or already show early signs of tumor cachexia is crucial for the establishment of effective cancer treatment. Comparative analysis of skeletal muscle biopsies taken from the abdomen of patients during indicated surgeries will be conducted. The patients will be allocated to the following study groups: a) Study group 1: Patients without cancer, b) Study group 2: Patients with solid tumors who did not perform physical training and c) Study group 3: Patients with solid tumors who executed physical training in form of WB-EMS. The investigation can help to understand skeletal muscle physiology under exercise and to get a better insight into the effects of physical training on early-stage muscle atrophy, both on cellular and molecular level. Initially, it is planned to identify the inflammation and nutrition status of the patients, and to determine skeletal muscle strength. It is anticipated to explore muscle protein composition, particularly myosin to actin ratio and their interaction. Biochemical analysis and the examination of the cellular ultra-structure should enhance the knowledge about the key mechanisms controlling the contractile apparatus of single muscle fibers in order to determine the quality of muscle force. Taken together, these investigations will help to better understand muscle atrophy in advanced cancer patients, and might support the development of targeted anti-cachectic therapies, that can be applied already in early phases of the tumor disease to significantly improve the patients' prognosis and their quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years
* Solid pancreatic, colorectal, esophageal, gastric and liver tumors under oncological treatment
* Karnofsky performance index between 50 and 100
* Loss of body weight (≥ 2 % and < 5 %, weight before the illness and at study entry)
* Distinct decrease in muscle force
* Indication for surgery proximal to the M. rectus abdominis
* Intervention Group must have an at least 8-week waiting period until the surgery (to conduct WB-EMS)

Exclusion Criteria:

* Participation in other nutrition or exercise intervention studies
* Study-independent exercise more than once a week
* Ingestion of anabolic or dietary supplements
* Occurrence of heavy cardio-vascular events
* Epilepsy and other severe neurological disorders
* Skin lesions in the area of the electrodes
* Conductive materials or electronical implants in the body (that do not allow electromyostimulation)
* Pregnancy
* Chronic diseases (e.g. HIV or Hepatitis C/D/E)
* Rejection of a muscle biopsy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 420 (Estimated)
Dates: Start 2017-05-31 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Differences in Myosin:Actin ratio | 8 weeks
  Myosin:Actin ratio in the muscle biopsies assessed by protein analysis via Western Blotting.
Differences in Myosin isoforms | 8 weeks
  The Myosin isoforms in the muscle biopsies will be determined by protein expression analysis via Western Blotting.
Differences in cellular ultra structures | 8 weeks
  Cellular ultra structures in the muscle biopsies will be examined using multi-photon microscopy.
Differences in Force development and Calcium 2+ sensitivity of single muscle fibers | 8 weeks
  Force development and Calcium 2+ sensitivity of single muscle fibers from the muscle biopsies will be assessed by in situ biomechanical recording.
Differences in activation of involved signaling pathways | 8 weeks
  Signaling pathways that regulate muscle atrophy will be analyzed by examining protein expression and modification (Western Blotting), and gene expression (quantitative PCR) in the muscle biopsies.

SECONDARY OUTCOMES:
Differences in inflammatory status | 0 week
  Pro-inflammatory cytokines
Differences in Nutritional risk | 0 week
  Nutritional Risk Screening-2002

CONTACTS AND LOCATIONS:
Locations (1):
- Hector-Center for Nutrition, Exercise and Sports, Erlangen, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No